CLINICAL TRIAL: NCT04443725
Title: Efficacy and Safety of Anti-hepatitis C Drugs in the Treatment of COVID-19
Brief Title: Efficacy and Safety of Anti HCV Drugs in the Treatment of COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamal Esmat, Professor of Endemic Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUKA-003
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine plus Sofosbuvir/Daclatasvir (Experimental): Hydroxychloroquine (hydroxychloroquine 400 mg by mouth twice daily for 1 day, then 200 mg by mouth twice daily for 14 days, Sofosbuvir 400 mg once daily for 14 days and daclatasvir 90 mg for 14 days
  Interventions: Drug: Hydroxychloroquine , Sofosbuvir, daclatasvir
- Standard of care (Active Comparator): Hydroxychloroquine 400 mg by mouth twice daily for 1 day, then 200 mg by mouth twice daily for 14 days
  Interventions: Drug: Standard of care treatment

INTERVENTIONS:
Drug: Hydroxychloroquine , Sofosbuvir, daclatasvir — Hydroxychloroquine (hydroxychloroquine 400 mg by mouth twice daily for 1 day, then 200 mg by mouth twice daily for 14 days (dose reductions for weight < 45 kg or GFR (glomerular filtration rate) <50ml/min) alone; as provided by the MOHP protocol), Sofosbuvir 400 mg once daily for 14 days and daclatasvir 90 mg for 14 days.
  Arms: Hydroxychloroquine plus Sofosbuvir/Daclatasvir
Drug: Standard of care treatment — Hydroxychloroquine (hydroxychloroquine 400 mg by mouth twice daily for 1 day, then 200 mg by mouth twice daily for 14 days (dose reductions for weight < 45 kg or GFR (glomerular filtration rate) <50ml/min) alone; as provided by the MOHP protocol),
  Arms: Standard of care

SUMMARY:
COVID 19 which started from a zoonotic transmission related to crowded markets was confirmed to have a high potential for transmission to close contacts on 20 January 2020 by the National Health Commission of China and it was announced as a pandemic by the WHO on 11 March 2020.

There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, conservation fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

Interestingly, sofosbuvir has recently been proposed as an antiviral for the SARS-CoV-2 based on the similarity between the replication mechanisms of the HCV and the coronaviruses.

Aim of the study is to assess the safety and efficacy of of the addition of HCV treatment to the standard regimen for the treatment of patients who are candidates to receive Hydroxy Chloroquine according to Egyptian MOHP protocol

DETAILED DESCRIPTION:
In December, 2019, an outbreak of pneumonia with unknown cause occurred in Wuhan city, the capital of Hubei province in China. On January 7th, the scientists succeeded to isolate a novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). WHO nominated it as coronavirus disease 2019 (COVID-19) in February, 2020.

COVID 19 which started from a zoonotic transmission related to crowded markets was confirmed to have a high potential for transmission to close contacts on 20 January 2020 by the National Health Commission of China and it was announced as a pandemic by the WHO on 11 March 2020.

SARS-CoV-2 infection have a wide clinical spectrum ranging between asymptomatic infection, mild upper respiratory tract symptoms, and severe viral pneumonia (fever, malaise, dry cough, shortness of breath, and respiratory distress) that may result in respiratory failure and finally death.

There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, conservation fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

For direct antiviral treatment of SARS-CoV-2, the China International Exchange and Promotive Association for Medical and Health Care (CPAM) recommended usage of lopinavir; ritonavir. Their recommendation was based on weak evidence from retrospective cohort, historically controlled studies, case reports, and case series reporting a clinical benefit of lopinavir; ritonavir in the management of other coronavirus infection [i.e., SARS-CoV 1 and Middle East respiratory syndrome coronavirus (MERS-CoV)] .

However, the first randomized clinical trial with lopinavir/ritonavir demonstrated no benefit over standard care in 199 hospitalized adults with severe COVID-19. There is no evidence to support the use of other antiretrovirals, including protease inhibitors; indeed, structural analysis demonstrates no darunavir binding to COVID-19 protease.

A group of Korean physicians experienced in SARS-CoV-2 infected patients' treatment developed recommendations for the treatment of COVID-19. According to them, antiviral medications lopinavir 400 mg; ritonavir 100 mg or chloroquine is considered to be used in older patients or patients with chronic health conditions and life threatening symptoms. If chloroquine is unavailable, hydroxychloroquine is recommended. Both of them have reported ability of inhibition of SARS-CoV-2 in vitro.

CPAM guidelines included them as they were associated with reduced progression of disease and decreased duration of symptoms. In an open-label study of 36 patients with COVID-19, use of hydroxychloroquine (200 mg three times per day for 10 days) was associated with a higher rate of undetectable SARS-CoV-2 RNA on nasopharyngeal specimens at day 6 compared with no specific treatment (70 versus 12.5 percent). In this study, the use of azithromycin in combination with hydroxychloroquine appeared to have additional benefit, but there are methodologic concerns about the control groups for the study, and the biologic basis for using azithromycin in this setting is unclear. In the United States, the FDA issued an emergency use authorization to allow the use of these agents in adolescents or adults hospitalized for COVID-19.

One of the studies done on SARS-COV-1 strongly suggested that using ribavirin as therapy should be reconsidered until further animal studies clarify the effects of ribavirin on cytokine and chemokine profiles during an infection and until ribavirin can be demonstrated to have a significant effect on reducing viral replication in vivo. Data from a molecular docking experiment using the SARS-CoV-2 RNA dependent RNA polymerase (RdRp) model identified tight binding of sofosbuvir and ribavirin to the coronavirus RdRp, thereby suggesting possible efficacy of sofosbuvir and ribavirin in treating the COVID-19 infection.

Chen et al. prepared the three-dimensional model of the SARS-CoV-2 (aka 2019-nCoV) 3C-like protease (3CL ) then performed virtual screening for purchasable drugs checking the actions, targets and side effects of the 16 candidates. Among these, we first noticed velpatasvir and ledipasvir, which are inhibitors of the NS5A protein of the hepatitis C virus (HCV). Both are marketed as approved drugs in combination with sofosbuvir, which is a prodrug nucleotide analogue inhibitor of RNA-dependent RNA polymerase (RdRp, or NS5B).

Interestingly, sofosbuvir has recently been proposed as an antiviral for the SARS-CoV-2 based on the similarity between the replication mechanisms of the HCV and the coronaviruses.

Based on this data the investigators suggest that these dual-component HCV drugs, Epclusa (velpatasvir/sofosbuvir) and Harvoni (ledipasvir/sofosbuvir), may be attractive candidates to repurpose because they may inhibit two coronaviral enzymes. A drug that can target two viral proteins substantially reduces the ability of the virus to develop resistance. These direct-acting antiviral drugs are also associated with very minimal side effects and are conveniently orally administered.

Aim of the study is to assess the safety and efficacy of the addition of HCV treatment to the standard regimen for the treatment of patients who are candidates to receive Hydroxy Chloroquine according to MOHP protocol.

ELIGIBILITY:
Inclusion Criteria:

* positive reverse-transcriptase-polymerase chain- reaction (RT-PCR) assay for SARS- CoV-2 in a respiratory tract sample

Exclusion Criteria:

* ● Known allergy or hypersensitivity to the used medications

  * Known severe liver disease (e.g., cirrhosis, with an alanine aminotransferase level >5× the upper limit of the normal range or an aspartate aminotransferase level >5× the upper limit of the normal range)
  * Use of medications that are contraindicated with the trial medications and that could not be replaced or stopped during the trial period
  * Pregnancy or breast-feeding or known active HCV infection, because of concerns about the development of resistance
  * History of bone marrow transplant
  * Known G6PD deficiency
  * Chronic hemodialysis or Glomerular Filtration Rate < 20ml/min
  * Psoriasis
  * Porphyria
  * Concomitant use of digitalis, flecainide, amiodarone, procainamide, or propafenone
  * Known history of long QT syndrome
  * Current known QTc>500 msec
  * Pregnant or nursing
  * Weight < 35kg
  * Seizure disorder
  * Patients receiving Amiodarone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Virological cure | 28 days
  virological cure using the triple therapy as compared to mono hydroxychloroquine treatment..

IPD SHARING:
Plan to Share IPD: Undecided